CLINICAL TRIAL: NCT00252889
Title: GSK - Doublet: A Phase I Study of Pegylated Liposomal Doxorubicin (Doxil) and Weekly Intravenous Topotecan in Patients With Advanced Solid Tumors
Brief Title: Doxil Topotecan Doublet Cancer Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: Johnson & Johnson (Industry); GlaxoSmithKline (Industry)
Responsible Party: Dr Gregory Masters MD Principal investigator, Christiana Care Health Services
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24062
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Small Cell Lung Cancer; Pancreatic Cancer; Head and Neck Cancer; Gastric Cancer; Esophageal Cancer
Keywords: Metastatic cancer; Metastatic gastric and esophagus adenocarcinoma; Unresectable pancreatic cancer; Unresectable head and neck cancer; Cancer of undetermined primary
MeSH Terms: conditions — Small Cell Lung Carcinoma; Pancreatic Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Neoplasm Metastasis; Adenocarcinoma Of Esophagus | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topotecan and pegylated doxorubicin — Doxil 40 mg/m2 day 1 and topotecan was to be escalated in cohorts of patients
  Other Names: Hycamptin Topoisomerase I inhibitor

SUMMARY:
The primary objective is to determine the nature and degree of the toxicity of weekly dosing of topotecan in escalating dose levels by cohorts of 3-6 patients in combination with a fixed dose of pegylated liposomal doxorubicin (Doxil).

The secondary objective is to determine the activity of weekly topotecan and pegylated liposomal doxorubicin in advanced solid tumors.

DETAILED DESCRIPTION:
Topotecan is a semisynthetic analogue of camptothecin. Like its parent compound camptothecin, topotecan is a specific inhibitor of topoisomerase-I. Topoisomerase-I facilitates DNA replication by inducing reversible single strand breaks thereby relieving the torsional strain which occurs ahead of the moving replication fork during DNA replication. Topotecan binds to the topoisomerase-I DNA complex and prevents relegation of the single strand breaks resulting in double strand DNA breaks. The cytotoxic action of topotecan is proportional to the cellular level of topoisomerase-I.

Doxorubicin is an anthracycline antibiotic which has a wide range of clinical activities. The mechanism of cytotoxicity and the exact intracellular target remains controversial. The bulk of intracellular drug is intranuclear much of which is intercalated in the DNA. Although DNA intercalation has been felt to be the principle cytotoxic mechanism, more recent evidence suggests inhibition of topoisomerase-II may play a more important role. Additionally, other cytotoxic actions including helicase inhibition have recently been noted. Pegylated liposomal doxorubicin (Doxil) is a polyethylene glycol pegylated liposomal encapsulation of doxorubicin. This results in an alteration of the pharmacokinetics in comparison to the parent compound. Specifically there is a prolonged circulation time, reduced clearance, a smaller volume of distribution, and limited uptake by the reticuloendothelial system. In animals using ovarian xenografts in nude mice, pegylated liposomal doxorubicin has resulted in a greater tumor to normal tissue drug uptake and an improved therapeutic index. Following phase I studies, Doxil has recently been studied in a phase II study of heavily pre-treated ovarian carcinoma patients with a response rate of 25.7%. This level of activity meets or exceeds other second-line agents currently available. In the recent phase II study, a dose of 50 mg/m2 every 3 weeks was utilized.

Topotecan given as 5 daily infusions is associated with significant myelosuppression and poor patient acceptance. Non hematologic toxicities are usually mild and not dose-limiting. Although the 5 day schedule can be inconvenient, the relative lack of acute toxicity still makes topotecan a good candidate for out-patient chemotherapy in selected patients. Although the impact of bone marrow suppression can be minimized by the use of cytokines, these 5 day regimens have required substantial dose reduction.

In view of the bone marrow toxicity seen with topotecan and the poor patient acceptance of a five day schedule, there has been interest in the development of an effective alternate treatment regimen using topotecan. Results from preclinical studies suggest that repeated administration of topotecan is necessary for its activity. A phase I study evaluating the safety and efficacy of weekly bolus topotecan as a second line agent in relapsed ovarian cancer resulted in a maximum tolerated dose of 5 mg/m2.

A phase II study in relapsed ovarian cancer supports the use of weekly topotecan at a dose of 3 - 4.0 mg/m2/week. Toxicities on this weekly regime have included, grade 3 or 4 neutropenia, anemia, thrombocytopenia, fatigue and GI toxicity, each occurred following less than 1% of treatments.

The combination of topoisomerase-I and topoisomerase-II inhibitors is an attractive strategy for cancer chemotherapy. A phase II study evaluated the combination of pegylated liposomal doxorubicin 30mg/m2/week with topotecan 1 mg/m2 IV for 5 consecutive days given every 28 days. Twelve patients with platinum resistant ovarian cancer were treated. Partial response was observed in three patients and four patients had stable disease of the ten patients evaluated for response. Toxicities included a higher percentage of bone marrow toxicity (grade III/IV neutropenia, grade III/IV thrombocytopenia) other toxicities included alopecia and diarrhea grade II/III. The authors concluded that the combination of topotecan and pegylated liposomal doxorubicin is active in the treatment of platinum resistant ovarian cancer. However, myelosuppression required dose reductions in nearly half the patients.

As mentioned earlier, a weekly regimen of topotecan has allowed for more convenient administration over more prolonged and more complex administration schedules. The current study will evaluate the tolerability of a weekly intravenous schedule of topotecan in combination with a standard dose of pegylated liposomal doxorubicin in advanced solid tumors. Due to the addition of the pegylated liposomal doxorubicin to a weekly schedule of topotecan, Pharmacokinetics data will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* ECOG functional status of 2 or better is required.
* The patient should be able to provide informed consent.
* Prior treatment with Doxil or topotecan is not permitted.
* Prior treatment with doxorubicin is permitted if the total dose was 350 mg/m2 or less. Prior treatment with epirubicin is permitted if the total dose was 560 mg/m2.
* Patients with controlled brain metastases will be considered eligible for therapy (i.e. metastases surgically removed; or irradiated metastases with stable neurologic function).
* Patients must have measurable disease (the presence of at least one measurable lesion).
* If previously irradiated lesions are to be used to measure response, documented growth of the lesions must have been observed following completion of radiation therapy.
* Patients must have a life expectancy of at least four weeks.
* Hematologic criteria: patients must have absolute neutrophil count (ANC) of 1200 or better; platelet count of 100,000/mm3 or better; hemoglobin (Hgb) ≥ 9.0g/dL.
* Hepatic criteria: bilirubin must be less than or equal to 1.7. SGOT, SGPT may be up to 2 x institutional upper limit of normal (ULN) but with the presence of liver metastasis the SGOT, SGPT may be up to 3 x institutional ULN.
* Serum creatinine must be < 1.5 mg/dl x ULN
* Patients with reproductive potential must use an adequate contraceptive method (e.g., abstinence, intrauterine device, oral contraceptives, barrier device with spermicide or surgical sterilization) during treatment and for three months after completing treatment.
* Patients must have a multigated acquisition (MUGA) scan or 2-d echocardiogram indicating an ejection fraction of ≥ 50% within 42 days prior to first dose of study drug. The method used at baseline must be used for later monitoring.

Exclusion Criteria:

* Patients with concurrent severe medical problems unrelated to malignancy, which would limit full compliance to the study or expose the patient to extreme risk with decreased life expectancy, are ineligible.
* Patients with previous or concomitant malignancy other than curatively treated carcinoma in situ of the cervix, basal cell or squamous cell carcinoma of the skin, or other primary cancer completely resected or treated within five years are ineligible. Exceptions are patients who have had tumors treated with no evidence of active disease who are felt by both the enrolling physician and the principal investigator (PI) to have a risk of relapse of less than 30%.
* Pregnant or lactating women.
* History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin hydrochloride (HCL) or the components of Doxil®.
* History of cardiac disease with New York Heart Association Class III or greater, or clinical evidence of congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-05; Primary Completion 2006-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Parameters of response: tumor measurement: Response Evaluation Criteria in Solid Tumors (RECIST) criteria | every other cycle
Survival is the observed length of life from the initiation of treatment to death or the date of last contact | follow up until death or loss of contact
Subjective parameters including ECOG performance status, specific symptoms, and side effects are graded according to standard Common Terminology Criteria for Adverse Events (CTCAE) v.30 criteria. | every cycle

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Guarino, M.D., Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health Services, Newark, Delaware, United States

REFERENCES:
- [Result] Masters GA, et. al., A Phase I Study of Pegylated Doxorubicin (DOX) and Weekly Topotecan (TOP) in Patients (pts) with Advanced Solid Tumors. ASCO Abstract, submitted 12/14/05.